CLINICAL TRIAL: NCT02361528
Title: A Double-Blind, Randomized, Placebo-controlled Multicenter Trial of GRanulocyte-Macrophage Colony-stimulating Factor Administration to Decrease ICU Acquired Infections in Sepsis-induced ImmunoDepression
Brief Title: GM-CSF to Decrease ICU Acquired Infections
Acronym: GRID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014.856
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Septic shock; Severe sepsis; GM-CSF; Immunosuppression; Hospital-acquired infections; ICU-acquired infections; HLA-DR; Monocytes
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leukine (Experimental): Sargramostim: Leukine (Genzyme USA), 125µg/m2 , once per day during 5 days, by subcutaneous route
  Interventions: Drug: Sargramostim: Leukine (Genzyme USA)
- placebo (Placebo Comparator): placebo, once per day during 5 days by subcutaneous route
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim: Leukine (Genzyme USA) — Leukine: 125 µg/m² daily, subcutaneously, for 5 days.
  Arms: Leukine
Drug: Placebo — placebo subcutaneously, for 5 days
  Arms: placebo

SUMMARY:
The concept of acquired immunodeficiency after a first severe infection in the ICU is widely described in the literature. There is a dual risk: increased mortality and increased secondary infections. Several approaches of immunostimulatory treatments have been proposed in the literature. The treatment proposed by this study consists of the administration of Granulocyte-macrophage colony-stimulating factor (GM-CSF), colony stimulating factor widely used particularly in the USA where it is marketed. A phase 2 clinical trial was conducted in Germany in 2009.

The main objective is to measure the incidence of ICU-acquired infections in 2 groups of patients treated by GM-CSF or placebo. ICU patients at risk are defined as surviving at D3 from a severe sepsis or septic shock and presenting a sepsis associated immunodepression. The detection of immunosuppressed patients will be achieved by measuring the HLA-DR (Human Leucocyte Antigen DR)with a threshold of less to 8000 sites.

Our hypothesis is that the number of secondary infections (primary endpoint) will be significantly reduced in the treated group.

ELIGIBILITY:
Inclusion Criteria:

ICU patients presenting a severe sepsis or a septic shock associated with a sepsis-induced immunosuppression.

1. - Severe sepsis OR septic shock defined by the association of: at least 2 criteria of Systemic Inflammation Response Syndrome (SIRS) a clinically or microbiologically defined infection and respectively at least one organ failure (level ≥ 2 in one organ failure of the SOFA score) OR the need of a vasopressor treatment (epinephrine or norepinephrine ≥ 0,25mg/kg/min for at least 6 hrs to maintain a systolic pressure ≥ 90 mmHg or a mean arterial pressure ≥ 65 mmHg).
2. - AND Sepsis-induced immunosuppression: reduced mHLA-DR levels (< 8,000 monoclonal antibodies (mAb) per cell at D3).

Exclusion Criteria:

1. - Therapeutic limitation
2. Evolutive hemopathy, neutropenia < 500/mm3, stemcell transplant
3. Solid tumor with on-going chemotherapy or radiotherapy
4. Human immunodeficiency virus (HIV) infection with CD 4 count < 200 cell/mm3
5. Immunosuppressive treatment (including corticosteroid at immunosuppressive dose : > 10 mg equivalent prednisolone and cumulative dose > 700 mg)
6. Primary immunodeficiency .
7. Extra corporeal circulation within one month
8. Recent cardio-pulmonary resuscitation (within the current clinical episode)
9. Patients admitted in ICU for extensive burns
10. Contraindications to sargramostim
11. Pregnant or lactating women
12. Participation to another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients presenting at least one ICU-acquired infection at D28 or ICU discharge. | At Day 28 or ICU discharge.
  ICU-acquired infections will be recorded in accordance with the definitions of the European CDC used in the French network of IAI surveillance Rea Raisin. An independent committee blinded to treatment group will ensure the classification of hospital-acquired infections.

SECONDARY OUTCOMES:
Incidence and incidence density of pneumonia, catheter related infections, and urinary tract infections | At Day 28 or ICU discharge.
Survival at D28, end of ICU and hospital stay, and at 1 year | At Day 28 or ICU discharge.
Organ failure free days | At Day 28 or ICU discharge.
Number of serious adverse events and number of patients having presented at least one serious adverse event. | At Day 28 or ICU discharge.

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU Amiens Hopital SUD, Amiens
  - CHU Estaing 1 place Lucie et Raymond Aubrac, Clermont-Ferrand
  - CHU Gabriel MONTPIED, Clermont-Ferrand
  - CHU de Grenoble- Hopital Michallon, Grenoble
  - CHU de Grenoble-Hopital Michallon, Grenoble
  - Hopital Edouard Herriot, Lyon
  - Hopital de la Croix Rousse, Lyon
  - APHM Hopital de la Timone, Marseille
  - CHU la Conception, Marseille
  - APHM Hopital Nord, Marseille
  - CHU Montpellier, Montpellier
  - Hopital Saint Eloi, Montpellier
  - CHU de Nantes, Nantes
  - PTMC CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU Hopital Nord, Saint-Etienne

REFERENCES:
- [Background] Vacheron CH, Lepape A, Venet F, Monneret G, Gueyffier F, Boutitie F, Vallin H, Schwebel C, Maucort-Boulch D, Friggeri A; GRID Study Group. Granulocyte-macrophage colony-stimulating factor (GM-CSF) in patients presenting sepsis-induced immunosuppression: The GRID randomized controlled trial. J Crit Care. 2023 Dec;78:154330. doi: 10.1016/j.jcrc.2023.154330. Epub 2023 May 31. PMID 37267804